CLINICAL TRIAL: NCT07275554
Title: Analysis of Methylomic Features and Prognostic Risk Prediction in Patients With Hepatitis B-related Acute-on-chronic Liver Failure
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202410-059-1
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: HBV Related Acute-on-chronic Liver Failure; HBV-related Liver Cirrhosis; HBV (Hepatitis B Virus)
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic hepatitis B
- Hepatitis B-related liver cirrhosis
- Hepatitis B-related acute-on-chronic liver failure

SUMMARY:
This study aims to investigate the methylomic features of patients with hepatitis B-related acute-on-chronic liver failure and establish and validate a prognostic risk prediction classification model. The findings are of significant importance for guiding clinical practice and improving patient prognosis. Additionally, a methylomics-based classifier model for liver failure will be developed for disease prognosis analysis and clinical assessment, with the potential to enhance the diagnostic efficiency of liver failure.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B was persistent hepatitis B surface antigen (HBsAg) seropositivity for more than six months.

Hepatitis B-related liver cirrhosis was diagnosed based on histological examination, typical features on ultrasound or radiological imaging, endoscopic findings of portal hypertension, and clinical history.

Hepatitis B-related acute-on-chronic liver failure meets the diagnostic criteria of the 2018 Asia-Pacific guidelines for the diagnosis and treatment of liver failure.Laboratory tests:Jaundice: Serum total bilirubin ≥ 85 µmol/L and coagulopathy [International Normalized Ratio (INR) ≥ 1.5 or Prothrombin Activity (PTA) < 40%].

Exclusion Criteria:

* co-infection with other hepatitis viruses; history of hepatocellular carcinoma or other malignancies; concomitant autoimmune liver disease; or insufficient clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with chronic hepatitis B, Hepatitis B-related liver cirrhosis, and Hepatitis B-related acute-on-chronic liver failure
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of Methylomic Features in Patients with Hepatitis B-Related Acute-on-Chronic Liver Failure | 48months

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China